CLINICAL TRIAL: NCT02428348
Title: EEG@HOME (Phase 3b of the Project, Interviews)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Project funding ended before Phase 3b could be completed.
Sponsor: University Hospital, Ghent (Other)
Collaborators: Pilipili NV (Industry); Imec (Industry)
Responsible Party: Principal Investigator, Neurologie, Prof. dr. Kristl Vonck, University Hospital, Ghent
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EC/2014/1283(2)
Record Dates: First submitted 2015-03-31; First posted 2015-04-28 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interview (Experimental): Interview of epilepsy patients and their family about their opinion on different EEG-cap models in development.
  Interventions: Other: Interview about prototype EEG-cap

INTERVENTIONS:
Other: Interview about prototype EEG-cap

SUMMARY:
The goal of this project is the development of an EEG-cap (min. 21 electrodes) with user-friendly active dry electrodes that meets the expectations of the users regarding comfort and esthetics, without losing sight of the functional and technical demands for recording high quality EEG signals. The purpose is to use the EEG-cap to investigate clinical neurological disorders (e.g. epilepsy). The EEG-cap could also be used at home so that hospital admission in the EMU can be avoided for some patients and an increasing number of patients can be examined.

Phase 3 of this Project will be divided into Phase 3a and Phase 3b.

In Phase 3b of the project epilepsy patients and their family will be interviewed about different EEG-cap models in development. This interview is anticipated to take approximately 1 hour.

Minimum 4 - maximum 20 epilepsy patients and their family will be interviewed.

The results of the interviews will be analysed by the design company pilipili nv.

ELIGIBILITY:
Inclusion Criteria:

* Epilepsy patient

Exclusion Criteria:

* No experience with EEG

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-01; Primary Completion 2015-04 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
User opinion (questionnaire) | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Ghent, Ghent, Belgium